CLINICAL TRIAL: NCT00903708
Title: A Phase I Dose-Escalation, Pharmacokinetic and Pharmacodynamic Evaluation of Intravenous LY2275796 in Patients With Advanced Cancer
Brief Title: LY2275796 in Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0770
Record Dates: First submitted 2009-05-15; First posted 2009-05-18 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Advanced Cancers
Keywords: Advanced Cancers; LY2275796; Eukaryotic initiation factor 4E; eIF-4E
MeSH Terms: interventions — LY 2275796

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY2275796 (Experimental)
  Interventions: Drug: LY2275796

INTERVENTIONS:
Drug: LY2275796 — 100 mg administered by vein as a loading dose daily over 3 days, and then as a maintenance dose weekly thereafter.

SUMMARY:
Primary Objective:

* To determine a recommended Phase 2 dose of LY2275796 that may be safely administered to patients with advanced cancer, with prospects for therapeutic biologic effects. This will require simultaneous:
* monitoring of toxicities & determination of maximal tolerated dose (MTD)
* detecting eIF-4E target inhibition in tumor
* pharmacokinetic measurements

Secondary Objectives:

* To estimate pharmacokinetic parameters of LY2275796 and explore pharmacokinetic/pharmacodynamic relationships
* To document any antitumor activity observed with LY2275796

DETAILED DESCRIPTION:
LY2275796 is designed to block the effect of a cancer-promoting gene called eIF-4E (eukaryotic initiation factor 4E).

Before you can receive the drug on this study, you will have what are called "screening tests." These tests will help the doctor decide if you are eligible to take part in the study. Your complete medical history will be recorded and you will have a physical exam. You will have an electrocardiogram (ECG -- a test that measures the electrical activity of the heart). You may also have x-rays, computed tomography (CT) scans, or magnetic resonance imaging, whichever imagining your doctor thinks is best to monitor the status of the disease.

Blood (about 3 tablespoons) will be drawn for routine tests and to measure how the drug moves around inside your body and effects your body. Your blood sample will also be tested for human immunodeficiency virus (HIV, the virus that causes AIDS), Hepatitis B, and Hepatitis C. If your test results show that you have HIV, Hepatitis B, or Hepatitis C, you will be notified and given information about counseling services. The results of your HIV, Hepatitis B, and Hepatitis C tests will be kept confidential and disclosed only as required by law. If you do not take these tests for Hepatitis B, Hepatitis C, or HIV, or if you test positive for any of these, you will not be eligible for this study. If there is more than a 2-week delay before beginning the study, these tests may need to be repeated. Within 3 days of receiving the study drug, women who are able to have children must have a negative blood pregnancy test.

If you are found eligible to take part in this study, LY2275796 will be given by an infusion into your vein over 3 days. This is called a loading dose of the study drug and the purpose is to make sure the tumor tissue gets enough of the study drug for it to target the disease. This dose will be given either as 3 separate 3-hour infusions by vein for 3 days in a row or as a nonstop infusion for 3 days (72 hours).

The way you receive the drug will be decided by your study doctor and the study sponsor. This decision will be based upon the dose of the study drug that you are to receive and on the information gathered from other participants who have already received the study drug. Whichever way you are to receive the study drug, you may have to stay in the hospital for the first 3 days. Days 1-7 will be considered Cycle 1 of this study.

After the first loading dose, you will continue to receive the study drug as a single, 3-hour infusion 1 time each week (this is called a maintenance dose). Maintenance doses will be given on Days 8, 15, and 22 as a single, 3-hour infusion. Days 8-28 will be defined as Cycle 2. All cycles beginning with Cycle 3 will be 28 days. In this study, different participants will receive different dose levels.

During the first 29 days of the study, you will give 16 blood samples (about 1 teaspoon each) for pharmacokinetic (PK) testing. PK testing measures the amount of study drug in the blood at different times. On Cycle 1 Day 1, blood will be drawn 3 hours after the drug is given. On Cycle 1 Day 3, blood will be drawn before the infusion, 1 hour after the drug is given, at the end of the infusion, and again 20 minutes, 1 hour, 3 hours, and between 4-6 hours after the end of the infusion. On Cycle 1 Days 4-6, blood will be drawn on 1 occasion. On Cycle 2 Day 8, blood will be drawn before the infusion, and at the end of the infusion. On Cycle 2 Day 15, blood will be drawn before the infusion, then again 3, 9, and 24 hours later. The last PK test will be drawn either at the time of your biopsy (Part B or C only) or before the next dose of study drug is given on Day 29.

These blood samples will be used to measure the amount of whole molecules of LY2275796 in your blood. However, smaller traces of LY2275796 may also be found. If there is a portion of blood left over, it will be used to detect these broken down molecules of the study drug in your blood, since testing for these traces may be an easier way to monitor the presence of LY2275796 in the blood and may be better a predictor of how long the drug effects the body.

To test the effect of the drug in your body, a blood sample will be drawn (about 1 tablespoon) at the beginning of all cycles before you take LY2275796.

During Part A of the study, 1 participant will be enrolled at a time. In this part, doses will be increased quickly, doubling the dose with each new participant enrolled. Participants will continue to be enrolled until blood tests show a certain amount of study drug or if a participant experiences an intolerable side effect. Part B will begin once this happens.

During Part B of the study, 3 participants will be given the same dose of the study drug. If all 3 participants tolerate the dose of study drug well, another 3 participants will enrolled at a higher dose. These dose increases will continue until tumor biopsies show that the drug is having the required effect on the cancer in all 3 participants at 1 dose (this is called the optimal biologic dose, or OBD). However, if 2 participants at 1 dose experience the same intolerable side effect, additional participants will be enrolled at slightly lower doses until the highest well tolerated dose is identified (this is called the maximum tolerated dose, or MTD) this will be the maximum tolerated dose (MTD). Once the MTD or OBD is found, Part C will begin.

Ten (10) participants will be enrolled in Part C. at the OBD or the MTD dose found in Part B.

If you are enrolled in Part B or Part C, you will have tumor biopsies. If you have tumors that can be felt under the skin, the biopsy may will be done after a local anesthetic is used to numb the skin. If the tumor is not detectable by touch, you would have the biopsy performed with the help of a CT scan or ultrasound. The first biopsy will be within 4 weeks before starting LY2275796. You will then have 1 more biopsy between 21-28 days after you start taking LY2275796. The first biopsy taken before you receive the study drug is to get a baseline evaluation of the tumor. The biopsy taken after you receive the study drug is to check the level of the study drug in the tumor and also to see if the drug is working in the cancer cells as it is expected to do.

On the days you receive the loading dose and weekly maintenance doses, your doctor will perform a physical exam. Blood (about 2 tablespoons) will be drawn to measure the effects of LY2275796 on your blood count, your blood chemistry, the ability of your blood to clot, liver and kidney function, and possibly to check your tumor. If needed, extra samples may be drawn to check blood levels of LY2275796.

You will be taken off study if you have intolerable side effects or the disease gets worse.

When you go off study, you will have a physical exam. Blood (about 2 tablespoons) will be drawn to measure the effects of LY2275796 on your blood count, your blood chemistry, the ability of your blood to clot, liver and kidney function, and possibly to check the tumor. You will have the same imaging studies that have been performed during the study to monitor the status of the disease.

You will also be required to visit your doctor about 30 days after your last dose of LY2275796 for follow-up tests. You will have a physical exam. Blood (about 2 tablespoons) will be drawn to measure the effects of LY2275796 on your blood count, your blood chemistry, the ability of your blood to clot, liver and kidney function, and possibly to check the tumor. You will have the same imaging studies that have been performed during the study to monitor the status of the disease. You also will be asked about any side effects you have experienced. If you have side effects, you will visit your doctor every 30 days until the side effect stops or you begin a new cancer treatment. If you have no side effects from the LY2275796, no further follow-up will be necessary for the study.

This is an investigational study. LY2275796 is not FDA approved or commercially available, and it has been authorized for use in research only. About 40 patients may participate in this multicenter study. About 20 patients will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of histologically or cytologically documented malignancy, including patients with treated, stable brain metastases. For Part A: Malignancy that is advanced and/or metastatic for which no proven therapy exists (for example, there is no comparable or satisfactory alternative drug or other therapy available to treat that stage of the disease). For Part B and C: Malignancy that is advanced and/or metastatic for which no proven therapy exists, and presents with disease that is amenable to serial measurement of pharmacodynamics by biopsy.
2. Male or female >/= 18 years of age
3. Written informed consent from the patient
4. Performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale
5. Patients must have discontinued all previous therapies for cancer, including chemotherapy, radiotherapy, or other investigational therapy for at least 4 weeks (2 weeks for palliative radiotherapy, 6 weeks for mitomycin C or nitrosoureas), prior to study enrollment and have recovered from the acute effects of therapy.
6. Patients are able to comply with the protocol requirements and are reliable and willing to make themselves available for the duration of the study and will abide by the research units policies and procedures.
7. Have adequate organ function including: Bone Marrow Reserve: Absolute neutrophil count (ANC) >/= 1.5 x 10^9/L prior to treatment, platelets >/= 100 x 10^9/L, hemoglobin >/= 9 g/dL; Hepatic: Bilirubin </= upper limits or normal (ULN), alanine transaminase (ALT) and aspartate transaminase (AST) </= 2.5 x ULN; Renal: Calculated creatinine clearance by Cockcroft-Gault formula >/= 50 ml/min; Coagulation: Activated prothrombin time (APTT) and prothrombin time (PT) less than or equal to the ULN.
8. Males and females with reproductive potential should use medically approved contraceptive precautions during the trial and for 3 months following the last dose of study drug.

Exclusion Criteria:

1. Patient with current hematological malignancies or bleeding diathesis
2. Serious pre-existing medical conditions at the discretion of the investigator
3. Major surgery within 4 weeks of study enrollment
4. Women who are pregnant or lactating
5. Symptomatic central nervous system (CNS) neoplasm. (Patients who have CNS neoplasms stable on steroid medication may be included.)
6. Concomitant anticancer therapy or anticoagulant therapy (with the exception of the use of heparinized saline to maintain the patency of central venous catheters).
7. Patients who require palliative radiotherapy at the time of study entry
8. Previous treatment with antisense therapies
9. Within 30 days of the initial dose of study drug, have received treatment with a drug that has not received regulatory approval for any indication
10. Presence of positive test results in HIV antibodies, Hepatitis B surface antigen, or Hepatitis C antibodies (Rationale: Correlative biologic studies entail aerosolization of biologic fluids. Researchers use Universal precautions and should be protected from HIV or Hepatitis viruses. However, robotic equipment handling specimens with high viral load would require purging and sterilization procedures that could damage the equipment or alter results for subsequent specimens. Patients lacking symptoms or signs of HIV or hepatitis have low viral loads so that screening for them is not necessary).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of LY2275796 | Dose toxicity with each loading dose (daily for 3 days) then weekly
  Maximum tolerated dose (MTD) defined as highest dose at which 0-1/6 patients experience Grade III toxicity with LY2275796 administered IV as a loading dose daily over 3 days, then as maintenance dose weekly.

CONTACTS AND LOCATIONS:
Overall Officials: David Hong, MD, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org